CLINICAL TRIAL: NCT04167436
Title: Fit for Surgery. Clinical Randomized Trial of Multimodal Prehabilitation Strategy in Patients With Colorectal Cancer.
Brief Title: Fit for Surgery. Multimodal Prehabilitation in Colorectal Cancer Patients
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zealand University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REG-040-2017
Record Dates: First submitted 2019-11-11; First posted 2019-11-18 (Actual); Last update posted 2022-03-03 (Actual); Status verified 2022-02

CONDITIONS: Colon Cancer; Rectal Cancer; Frailty
Keywords: Prehabilitation; Colon cancer; WHO performance status; Rectal cancer; Exercise; Nutritional supplement
MeSH Terms: conditions — Colonic Neoplasms; Rectal Neoplasms; Frailty; Motor Activity | interventions — Preoperative Exercise

STUDY DESIGN:
Intervention Model Description: Randomized Clinical Trial with an intervention arm and a standard of care arm.
Who Masked: Outcomes Assessor
Masking Description: Due to the nature of the interventions neither participant, care provider or investigator is blinded. Outcome assessor of primary outcomes are blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Prehabilitation (Experimental): Patients receive multi-modal prehabilitation with exercise three times weekly, protein supplements, vitamin supplements, dietitian consultation and medical optimization prior to surgery. A minimum of four weeks.
  Interventions: Other: Prehabilitation
- Standard of Care (No Intervention): Receives standard of care

INTERVENTIONS:
Other: Prehabilitation — A minimum of four weeks of prehabilitation with exercise three times a week, protein and vitamin supplements, dietitian consultation and medical optimization prior to surgery.
  Arms: Prehabilitation

SUMMARY:
Randomized clinical trial of multimodal prehabilitation in vulnerable patients with colon or rectal cancer prior to surgery.

DETAILED DESCRIPTION:
Fit for surgery is a randomized clinical trial of multimodal prehabilitation prior to colon or rectal cancer surgery. Participants will either receive

The study is a part of the PREHAB study which is performed in collaboration with international centers.

The full protocol are published BMC Cancer. 2019 Jan 22;19(1):98. doi: 10.1186/s12885-018-5232-6.

ELIGIBILITY:
Inclusion Criteria:

* Undergoing elective colorectal cancer surgery
* WHO performance status I and II
* Signed consent

Exclusion Criteria:

* Known metastatic disease
* Unable to perform baseline test or basic training e.g. paralytic or completely immobilized patients, orthopedic impairments.
* ASA 4 or 5 (American Society of Anesthesiologist Classification)
* Neoadjuvant chemo- or radiation therapy
* Renal failure III B or higher
* Illiteracy or unable to write or understand Danish
* Cognitive disabilities, which affects adherence e.g. severe dementia (MMSE score ≤17).
* Withdrawal of consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2019-05-01 (Actual); Primary Completion 2022-05-01 (Estimated); Study Completion 2022-08-01 (Estimated)

PRIMARY OUTCOMES:
Quality of Recovery 15 | 3 days after surgery
  Difference in postoperative recovery between baseline and within 3 days after surgery. The cumulative score ranges from 0-150, with a higher value indicating a better outcome
Changes in physical fitness prior to surgery | Baseline, prior to surgery and 30 days after surgery
  Changes in VO2 max between baseline and prior to surgery
Complications | 30 days after surgery
  Complications measured by the comprehensive complication index. The score ranges from 0-100 with with a higher value indicating a worse outcome.
Changes in immunological function | Blood work taken at baseline, prior to surgery, three days after surgery and four weeks after surgery. Tumor from resectionspecimen
  Changes in immunological function measured by nanostring in blood and tumor (in the invasive front)

SECONDARY OUTCOMES:
Disease specific quality of life - EORTC c30 | the day prior to surgery, 30 days after surgery, 60 days after surgery and one year after surgery
  European Organisation for Research and Treatment of Cancer Questionaire c 30 (EORTC c30). The EORTC c30 contains 6 domains which will each be assessed for mean changes in their cumulative score. The domains are physical function, role function, emotional function, pain, fatigue and global health. A higher value indicating a worse outcome
Disease specfic quality of life - EORTC c29 | the day prior to surgery, 30 days after surgery, 60 days after surgery and one year after surgery
  European Organisation for Research and Treatment of Cancer Questionaire c 29 (EORTC). The questionnaire contains 29 items, with a 4 point Likert scale for symptoms and 7 point Likert scale for quality of life and global health. For the 4 point Likert scale the higher the score the worse the outcome. For the 7 point likert scale higher values indicating a better outcome. Analysis will be performed for changes in individual symptoms and cumulative aggregation of scores will not be performed.
Overall quality of life - SF-36 | the day prior to surgery, 30 days after surgery, 60 days after surgery and one year after surgery
  Short Form 36 question (SF-36) health questionnaire. The questionnaire contains eight domains: physical functioning, pain, limitations due to physical health problems, limitations due to personal or emotional problems, emotional well-being, social functioning, fatigue, and general health perceptions. Scores for each domain range from 0 to 100 and the analysis will be performed as mean difference between baseline and the following time frame. A higher value indicating a better outcome.
Psychological health - Depression - PHQ-9 | the day prior to surgery,30 days after surgery, 60 days after surgery and one year after surgery
  Patient Health Questionnaire 9 (PHQ-9) Depression test. The PHQ-9 have a maximum of 27 points and a minimum of 0. The outcome is point change between baseline and following time frame. A higher value indicating a worse outcome
Psychological health - General anxiety - GAD-7 | the day prior to surgery, 30 days after surgery, 60 days after surgery and one year after surgery
  General Anxiety Disorder 7-item (GAD-7). The questionnaire have a maximum of 21 points and a minium of 0. The outcome is the point change between baselin and the following time frame. A higher value indicating a worse outcome
Physical function (6-MWT) | The day prior to surgery, 30 days after surgery, and 60 days after surgery
  6-Minutes walk test. Measures how far the participant can walk in 6 minutes measured in meters
Physical function (STS) | The day prior to surgery, 30 days after surgery, and 60 days after surgery.
  Sit-to-stand test. Test of how many times the patient can rise from a chair in 30 seconds.
Physical function (Stair climb test) | The day prior to surgery, 30 days after surgery, and 60 days after surgery
  Stair climb test will be measured as the number of steps (17 mc in height) the paitent can rise in 30 secounds.
Physical function (Leg extension test) | The day prior to surgery, 30 days after surgery, and 60 days after surgery
  Leg extension test will be measured by fixed dynaometer in newtons three times on each leg and the maximum for each leg used for analysis.
Physical function (Hand grip strength) | The day prior to surgery, 30 days after surgery, and 60 days after surgery
  Hand grip strength measured by hand-held dynanometer in kilograms. Measured 3 times on each hand and will use the maximum obtained.
Nutritional status | The day prior to surgery, 30 days after surgery, and 60 days after surgery
  Increase/decrease in total body weight in percent.
Remission and cancer free survival | 5 years
  Remission and cancer free survival

CONTACTS AND LOCATIONS:
Locations (2):
- Denmark (2):
  - Zealand University Hospital, Køge, Danmark
  - Slagelse Hospital, Slagelse, Danmark

REFERENCES:
- [Derived] Bojesen RD, Dalton SO, Skou ST, Jorgensen LB, Walker LR, Eriksen JR, Grube C, Justesen TF, Johansen C, Slooter G, Carli F, Gogenur I. Preoperative multimodal prehabilitation before elective colorectal cancer surgery in patients with WHO performance status I or II: randomized clinical trial. BJS Open. 2023 Nov 1;7(6):zrad134. doi: 10.1093/bjsopen/zrad134. PMID 38060453
- [Derived] Molenaar CJ, van Rooijen SJ, Fokkenrood HJ, Roumen RM, Janssen L, Slooter GD. Prehabilitation versus no prehabilitation to improve functional capacity, reduce postoperative complications and improve quality of life in colorectal cancer surgery. Cochrane Database Syst Rev. 2023 May 10;5(5):CD013259. doi: 10.1002/14651858.CD013259.pub3. PMID 37162250
- [Derived] Molenaar CJ, van Rooijen SJ, Fokkenrood HJ, Roumen RM, Janssen L, Slooter GD. Prehabilitation versus no prehabilitation to improve functional capacity, reduce postoperative complications and improve quality of life in colorectal cancer surgery. Cochrane Database Syst Rev. 2022 May 19;5(5):CD013259. doi: 10.1002/14651858.CD013259.pub2. PMID 35588252
- [Derived] Bojesen RD, Jorgensen LB, Grube C, Skou ST, Johansen C, Dalton SO, Gogenur I. Fit for Surgery-feasibility of short-course multimodal individualized prehabilitation in high-risk frail colon cancer patients prior to surgery. Pilot Feasibility Stud. 2022 Jan 21;8(1):11. doi: 10.1186/s40814-022-00967-8. PMID 35063042